CLINICAL TRIAL: NCT04046757
Title: Strategy for Transfer to Emergency Head And Neck (UTEC) of Stroke Alerts With Suspicion of Large Vessel Occlusion for Mechanical Thrombectomy in the Languedoc Roussillon Region
Brief Title: Regional Strategy for Transfer for Mechanical Thrombectomy
Acronym: START
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0378
Record Dates: First submitted 2019-06-07; First posted 2019-08-06 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Stroke; Ischemic; Large Vessel Occlusion
Keywords: Ischemic stroke; Mechanical Thrombectomy
MeSH Terms: conditions — Stroke; Ischemia; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mechanical thrombectomy — Neuroradiological endovascular treatment

SUMMARY:
A mono-centre observational study with the aim of compare clinical outcome at 3 month on patients admitted with recent cerebral infarct and intracranial large vessel occlusion in the anterior circulation who are eligible for mechanical thrombectomy in three different position : Patients admitted first in the Comprehensive Stroke Center of Montpellier, those transferred after Proximity Stroke Unit or prehospital bypass for patients with high suspicion of large vessel occlusion.to the Comprehensive Stroke Center of Montpellier

DETAILED DESCRIPTION:
Multiple RCT has recently proved the superiority of mechanical thrombectomy compared to the best medical therapy (BMT) on patients with recent cerebral infarct and anterior circulation intracranial large vessel occlusion.

In the Occitanie-Est region (ex Languedoc Roussillon), comprising 6 Stroke Unit, only the Comprehensive Stroke Unit of the CHU de Montpellier has a centre of interventional neuroradiology (NRI) that can perform mechanical thrombectomy.

Patients suspected of stroke are referred to the nearest SU, then the candidates for thrombectomy, are transferred secondarily to the Stroke Center in Montpellier.

Currently, there is no evidence that an initial management in a proximity stroke unit and a secondary transfer for a mechanical thrombectomy is associated with a loss of chance for patients, compared to patients initially treated at the Stroke Center regional reference.

The objective of the study is to compare clinical outcome on patients admitted first in the Comprehensive Stroke Center of Montpellier those transferred after Proximity Stroke Unit or directly admitted when high suspicion of large vessel occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patient, admitted to the Emergency Department Head and Neck of the CHU de Montpellier, over 18 years old, without limit of upper age
2. With TIA or cerebral infarction (confirmed by brain imaging (MRI or CT scan), acute (Time of stroke symptoms or discovery of patient ≤ 12 h)
3. With anterior circulation intracranial large vessel occlusion (M1, T or proximal M2), confirmed by arterial imaging (magnetic resonance angiography-MRA- or angioscanner)
4. No objection of the patient or their representative to being included in the cohort

Exclusion Criteria:

1. Patient with severe intercurrent pathology impacting the short-term vital prognosis and making follow-up impossible
2. Predictable impossibility of patient follow-up

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute cerebral infarct in the arterial circulation with large vessel occlusion
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Score (mRS) | 3 months
  Good functional outcome ( defined by a Modified Rankin Scale of 0-2, 3 months after stroke onset Modified Rankin scale . Range 0 (asymptomatic) to 6 (death)
  * Good outcome : 0 to 2
  * Disability : 3 to 5
  * Bad outcome : 5 and 6

SECONDARY OUTCOMES:
Incidence of mechanical thrombectomy treatment | 24 hours
  Safety of medical complication
  Complications of mechanical thrombectomy :
  * Vessel perforation
  * Intramural Arterial dissection
  * Symptomatic Intracerebral hemorrhage
  * embolization to a new territory
Clinical evolution at 24 hours | 24 hours
  NIHSS scale and NIHSS scale variation between the inclusion at 24 hours
  National Institutes of Health Stroke Scale (NIHSS). Range 0-42. Neurological severity score at the acute phase :
  * Minor stroke : 0 to 5
  * Moderate stroke 6 to 20
  * Severe stroke up to 21
Clinical evolution 7 days | 7 days
  NIHSS scale and NIHSS scale variation between the inclusion at 7 days
  National Institutes of Health Stroke Scale (NIHSS). Range 0-42. Neurological severity score at the acute phase :
  * Minor stroke : 0 to 5
  * Moderate stroke 6 to 20
  * Severe stroke up to 21
Proportion of patients having had mechanical trombectomy (and/or intravenous thrombolysis) amongst patient cohort. | 24 hours
  Number of patients having had mechanical trombectomy (and/or intravenous thrombolysis) amongst patient cohort.
Symptomatic Intracerebral Haemorrhage | 24 hours
  symptomatic Intracerebral Haemorrhage on cerebral imaging at 24 hours
Arterial Recanalisation with TICI score | post-act / 24 hours
  Quality of revascularization after mechanical thrombectomy : immediate post-Mechanical-Trombectomy evaluation for patient having had mechanical thrombectomy and at 24 hours for all patient cohort.
  TICI score (Thrombolysis In Cerebral Infarction grading system) describe the quality of revascularization after mechanical thrombectomy (Grade 0 for no perfusion at 3 for Complete perfusion)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline ARQUIZAN, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Gui De Chauliac Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided